CLINICAL TRIAL: NCT04537169
Title: Clinical Significance of Whitnall Ligament Structure in Patients With Congenital Ptosis
Brief Title: Clinical Significance of Whitnall Ligament Structure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Sameh S. Mandour, Assistant Professor of Ophthalmology, Menoufia University
Other Study IDs: OPHTH2/2020
Record Dates: First submitted 2020-08-18; First posted 2020-09-03 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-08

CONDITIONS: Congenital Ptosis
Keywords: Whitnall ligament; congenital ptosis; levator resection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Mild congenital ptosis: children with mild congenital ptosis
  Interventions: Procedure: Levator resection
- Moderate congenital ptosis: children with moderate congenital ptosis
  Interventions: Procedure: Levator resection
- Severe congenital ptosis: children with severe congenital ptosis
  Interventions: Procedure: Levator resection

INTERVENTIONS:
Procedure: Levator resection — Eyelid crease incision Dissection of the levator aponeurosis to the level of Whitnall ligament. Assessment of the structure of Whitnal ligament. Resection of a calculated part of the aponsurosis. re-attachment of the aponeurosis to the tarsus Incision closure with crease formation

SUMMARY:
Prospective clincal study to relate the structure of Whitnall ligament in cases of congenital ptosis to the severety of ptosis and the postoperative results.

DETAILED DESCRIPTION:
The study will be a prospective obsevational study. It will include patients (2-16 years old) who will undergo levator resection for simple congenital ptosis correction in Ophthalmology Department of Menoufia University Hospital.

Patients will be divided into 3 groups, 15 patients in each. Group I for mild ptosis, Group II for moderate ptosis Group 3 for severe ptosis.

Exclusion criteria included any patients with previous ptosis or any eyelid surgery and patients with a non congenital ptosis.

Patients included in the study well be informed about the research and the surgical maneuver which will be used with full discussion of all details regarding the postoperative follow up and the potential complications. A written consent in Arabic will then be taken from the parents of the patients

Preoperative assessment will include Complete ophthalmological examination including; Margin to Reflex Distance 1 (MRD1), Vertical Fissure Height (VFH), Levator function (LF), and eyelid crease shape and position.

Intraoperative assessment will include Whitnall ligament structure assessment including:

* The level (the length from the insertion of the levator aponeurosis to Whitnall's ligament)
* Shape (definite band-like, weak string, undifferentiated)
* Tightness.

Postoperative assessment will be on scheduled visits at first week, one month, 3 months and 6 months postoperatively and will include MRD1, VFH, LF, and lagophthalmos measurements

Results will be documented and tabulated and statistically managed.

ELIGIBILITY:
Inclusion Criteria:

* Congenital ptosis

Exclusion Criteria:

* Previous ptosis surgery
* Non congenital ptosis

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Caucasian
Study Population: patients with congenital ptosis
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2020-08-20 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Success of levator resection in relation to structure of Whitnall ligament | An average of 1 year
  Relating the structure of the ligament with the degree of severity of ptosis by studying its position, shape and tightness in all cases during surgery

CONTACTS AND LOCATIONS:
Overall Officials: Richard C Allen, Study Chair — Department of Ophthalmology, Cullen Eye Institute,
Locations (1):
- Ophthalmology Department, Menoufia University Hospital, Shibīn al Kawm, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: No